CLINICAL TRIAL: NCT04014257
Title: A Phase 1, Open-label, Dose-escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of NOV1601(CHC2014) in Adult Subjects With Solid Organ Malignancies
Brief Title: A Phase 1 Study of NOV1601(CHC2014) in Adult Subjects With Solid Organ Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Collaborators: CMG Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV160101-101
Record Dates: First submitted 2019-07-02; First posted 2019-07-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Phase 1; Solid Tumor, Adult
Keywords: tropomyosin receptor kinase; Solid organ malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOV1601(CHC2014) (Experimental): a highly selective pan-TRK(tropomyosin receptor kinase) inhibitor targeting tropomyosin receptor kinase A(TRKA), tropomyosin receptor kinase B(TRKB), and tropomyosin receptor kinase C(TRKC)
  Interventions: Drug: NOV1601(CHC2014)

INTERVENTIONS:
Drug: NOV1601(CHC2014) — a highly selective pan-TRK(tropomyosin receptor kinase) inhibitor targeting tropomyosin receptor kinase A (TRKA), tropomyosin receptor kinase B(TRKB), and tropomyosin receptor kinase C(TRKC)

SUMMARY:
This study is a first-in-human (FIH) study which is required to understand the PK characteristics, MTD, and safety profile of NOV1601(CHC2014) in subjects with solid organ malignancies.

DETAILED DESCRIPTION:
This is the first-in-human, Phase 1, open-label, multicenter, dose-escalation study to investigate the safety, tolerability, PK, and clinical activity of NOV1601(CHC2014) in subjects with solid organ malignancies. The primary goal of the study is to determine the RP2D of NOV1601(CHC2014) in adult subjects with solid organ malignancies.

Dose escalation will follow a 3+3 design and will be based on prior cohort review. There will be 2 branches of the dosing schedule, once a day(QD) and twice daily(BID).

ELIGIBILITY:
Inclusion Criteria(partial):

* Pathological confirmation of malignancy and evidence of metastatic or surgically unresectable disease
* At least one evaluable or measurable lesion should be present and identified according to Response Evaluation Criteria in Solid Tumors(RECIST) version 1.1 or Response Assessment in Neuro-Oncology(RANO)
* Relapse after or refractory to systemic drug therapy to malignancy, at least one regimen of cytotoxic chemotherapy, kinase inhibitors including tyrosine kinase inhibitors or immunotherapy which is considered as standard of care if there is no standard regimen recommended, then no experience of systemic drug therapy is acceptable
* Patients with primary central nervous system(CNS) tumors or metastasis, if they have been neurologically stable

  * Symptoms should be under control by stable dose of glucocorticoids and analgesic drugs for symptom control at least 2 weeks prior to starting the treatment
  * Stable dose of glucocorticoids and analgesic drugs for symptom control should be maintained throughout the study
  * Subjects should be off from radiotherapy for at least 14 days prior to the start of study treatment(C1D1) without symptom aggravation

Exclusion Criteria(partial):

* Prior high-dose chemotherapy requiring hematopoietic stem cell transplantation
* History or evidence of suspicious leptomeningeal disease
* Previous surgery of gastrectomy, gastrostomy or any medical condition which interferes with oral ingestion of capsule
* Indwelling percutaneous drainage of bile and chest tube
* Evidence of or suspicious symptomatic spinal cord compression, unless appropriately treated and neurologically stable off glucocorticoid for at least 2 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
the recommended Phase 2 dose(RP2D) or the maximum tolerated dose(MTD) of NOV1601 | Subjects will be treated and observed for dose-limiting toxicity(DLT) through the end of the first cycle (Days 1-28).
  MTD will be the RP2D, based on the pharmacokinetic(PK) profiles and safety profiles as assessed by the Safety Monitoring Committee (SMC).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events(TEAE) and serious adverse events(SAE) | Maximum 2 years
  Each adverse event will be coded using the Medical Dictionary for Regulatory Activities(version 20.0) classification system. The severity of the toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wan Kim, MD, PhD, Principal Investigator — Seoul National University Hospital; Tak Yun, MD, PhD, Principal Investigator — National Cancer Center; Sang-Joon Shin, MD, PhD, Principal Investigator — Severance Hospital; Yong-Wha Moon, MD, PhD, Principal Investigator — CHA Bundang Medical Center
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul